CLINICAL TRIAL: NCT00156364
Title: "Ii-Pancreas Transplantation in Man", "Long Term Effects of Cyclosporine (CSA) and Tacrolimus (FK506) on Renal Structure and Function", "Studies of the Renal Interstitium Type I Diabetic Patients",
Brief Title: Studies of Organ Transplantation in Animals and Man
Status: Completed | Type: Observational
Sponsor: Michael Mauer, MD (Individual)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: University of Minnesota (Other)
Other Study IDs: 8107M00116; NIH 2P01-DK13083-38 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Diabetes Mellitus
Keywords: Diabetic Nephropathy; Kidney Transplant; Pancreas Transplant; Renal Interstitium; Diabetes Mellitus; Cyclosporine; Tacrolimus
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin Fibroblasts, Plasma and Serum samples, Urine samples, kidney biopsy culture samples.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A. To study the effects of pancreas transplantation (PT) on the structural abnormalities of diabetic nephropathy (DN) in patients with type 1 (insulin-dependent) diabetes mellitus (type 1 D). These studies will address the influence of long-term normoglycemia on two stages of diabetic renal disease.

Due to the difficulties encountered for recruitment of patients to agree to undergo a GFR and a native kidney biopsy in conjunction with their clinical evaluation visit for transplant, we are now focusing efforts on obtaining skin biopsies previous to transplant, and then at regular intervals (3, 6, and 9 months, and yearly) following a successful transplantation.

* Pancreas Transplantation Alone (PTA). To determine, at 5, 10, and 15 years after PTA, the effects of normoglycemia on the established lesions of DN in the long-term type 1 D patients' own kidneys.
* Islet Transplantation Alone (ITA). To determine, at 5 years after ITA, the effects of normoglycemia on the early lesions of DN in type 1 D patients' own kidneys.
* Pancreas Transplantation after Kidney Transplantation (PAK). To determine at 5-10 years the effects of normoglycemia on the early structural lesions of DN in kidneys transplanted some years earlier into type 1 D recipients.

Hypothesis: The benefits of PT on the early glomerular lesions of DN will be demonstrable after 5 years in kidneys exposed to diabetes for a short duration, while in patients with long-standing type 1 D and more advanced glomerular DN lesions, longer exposure to euglycemia is necessary to demonstrate arrest or regression of the lesions.

DETAILED DESCRIPTION:
These continuation studies focus on large pancreas (PTx) and kidney (KTx) transplant populations of type 1 diabetic (D) patients (pts) in order to better understand diabetic nephropathy (DN), the leading cause of renal failure. Objectives are: (a) to determine whether PTx can more readily arrest or reverse the early vs. the more established lesions of DN; (b) to continue studies of renal structural-functional relationships in DN, with emphasis on the multifaceted pathologic DN lesions, including glomerular, vascular, interstitial lesions and glomerular-tubular connections; (c) to continue studies of DN natural history and the role of renal biopsy in predicting outcome; (d) to quantitate and understand the basis of atubular glomeruli (AG) in DN; (e) to elucidate glomerular (glom) epithelial cell abnormalities in DN; (f) to study the glom extracellular matrix abnormalities of DN; (g) to study the recurrence of DN in the KTx; (h) to study the molecular/genetic basis of DN and develop cellular markers of DN risk; (i) to determine the long-term (10-15 yr) structural consequences of cyclosporine (CSA) on the native kidneys of PTx recipients; and (j) to determine the shorter-term (5 yr) consequences of Prograf on the native kidneys of PTx recipients and compare these with those seen after 5 years of CSA treatment. Together, these studies will help to elucidate the pathogenesis and natural history of DN, unravel some of the molecular and genetic aspects of this disease, describe the dynamics of DN reversal in PTx pts, and recurrence in KTx pts and expand our knowledge of the nephrotoxic effects of calcinosis inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Pancreas Transplantation. The patients considered for recruitment are those being evaluated for pancreas transplant alone or pancreas transplant after kidney transplantation in IDDM patients at the University of Minnesota (U of M). The consent forms have been approved by the Institutional Review Board at the University of Minnesota and the transplant coordinators responsible for interacting with patients have continuously utilized these consent forms in the recruitment process.
2. Long-Term Post Kidney Transplant IDDM Patients. These patients are recruited by a study coordinator working directly with the PI and also use consent forms approved by the Institutional Review Board at the University of Minnesota.

Exclusion Criteria:

Pancreas Transplantation Alone

1. Serum creatinine >1.5 mg/dl or CCr <50 ml/min/1.73M2, as kidneys in such IDDM patients are approaching end stage renal disease and are not readily amenable to morphometric analysis.
2. Solitary kidneys or evidence of unilateral renal disease, based upon significant discrepancies in renal size by ultrasound.
3. Evidence of other important kidney disease by history, ultrasound, or baseline biopsy.
4. Other chronic diseases or conditions, in addition to IDDM, such as cystic fibrosis, serious mental illness, severe mental retardation, etc.
5. Pregnancy. Pregnancy tests will be performed on all eligible females of child-bearing age, and pregnant women will be excluded. Patients will again be eligible 3 months after completion of pregnancy.

Pancreas Transplantation After Kidney Transplantation

1. Serum creatinine >2 mg/dl; a higher value is accepted than for native kidney patients since patients have a single kidney and are receiving CSA or FK506.
2. Moderate to severe chronic rejection on baseline biopsy.
3. Evidence of other important kidney disease by history, ultrasound, or baseline biopsy.
4. Other chronic diseases or conditions, in addition to IDDM, such as cystic fibrosis, serious mental illness, severe mental retardation, etc.
5. Pregnancy. Pregnancy tests will be performed on all eligible females of child-bearing age, and pregnant women will be excluded. Patients will again be eligible 3 months after completion of pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: This is not a study that recruits from the general population. This study is selectively offered to eligible patients who are scheduled for a Pre-pancreas Transplant evaluation visit at the University of Minnesota Medical Center, Fairview Transplant Center. If interested in learning more, contact the Transplant Center for more information.
Sampling Method: Probability Sample
Enrollment: 655 (Actual)
Dates: Start 1981-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Structural-functional relationships in diabetic nephropathy through detailed quantitative studies of Podocytes. | baseline through follow-up biopsy
  structural-functional relationships in diabetic nephropathy through detailed quantitative studies of podocytes, including cell number, shape and attachment using innovative approaches including quantitative immunoelectron microscopy and 3-dimensional high resolution electron microscopy. We will also study relationship between podocyte and glomerulotubular junction abnormalities.

SECONDARY OUTCOMES:
We will continue our study the natural history of diabetic nephropathy. | Baseline through follow up visits
  We will study the structural parameters associated with urinary albumin excretion and determine which structural parameters are predictors of developing diabetic nephropathy.

OTHER OUTCOMES:
We have compared the development of calcineurin lesions in the native kidneys of 14 tacrolimus- and 12 calcineurin-treated pancreas transplant alone recipients cured of type 1 diabetes. | Baseline through follow-up
  To avoid the pitfalls of renal allograft studies, including rejection and disease recurrence, we compared the development of calcineurin lesions in the native kidneys of 14 tacrolimus- and 12 calcineurin-treated pancreas transplant alone recipients cured of type 1 diabetes.
  Results: The cyclosporine and tacrolimus groups had, respectively, on average, 33% versus 44% decline in GFR (ns), 27% versus 29% increase in cortical interstitial fractional volume (ns), 245% versus 347% increase in the fractional volume of cortical tubules that were atrophic (ns), and 291% versus 392% increase in the percent of globally sclerotic glomeruli (ns). Arteriolar hyalinosis did not change significantly in either group.

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Mauer, MD, Principal Investigator — Pediatric Nephrology, University of Minnesota; Arthur J Matas, MD, Study Director — University of MN, School of Medicine, Dept of Surgery
Locations (1):
- Universtity of Minnesota, Department of Pediatric Nephrology, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Moriya T, Groppoli TJ, Kim Y, Mauer M. Quantitative immunoelectron microscopy of type VI collagen in glomeruli in type I diabetic patients. Kidney Int. 2001 Jan;59(1):317-23. doi: 10.1046/j.1523-1755.2001.00493.x. PMID 11135085
- [Background] Sutherland DE, Gruessner RW, Dunn DL, Matas AJ, Humar A, Kandaswamy R, Mauer SM, Kennedy WR, Goetz FC, Robertson RP, Gruessner AC, Najarian JS. Lessons learned from more than 1,000 pancreas transplants at a single institution. Ann Surg. 2001 Apr;233(4):463-501. doi: 10.1097/00000658-200104000-00003. PMID 11303130
- [Background] Caramori ML, Kim Y, Huang C, Fish AJ, Rich SS, Miller ME, Russell G, Mauer M. Cellular basis of diabetic nephropathy: 1. Study design and renal structural-functional relationships in patients with long-standing type 1 diabetes. Diabetes. 2002 Feb;51(2):506-13. doi: 10.2337/diabetes.51.2.506. PMID 11812762
- [Background] Katz A, Caramori ML, Sisson-Ross S, Groppoli T, Basgen JM, Mauer M. An increase in the cell component of the cortical interstitium antedates interstitial fibrosis in type 1 diabetic patients. Kidney Int. 2002 Jun;61(6):2058-66. doi: 10.1046/j.1523-1755.2002.00370.x. PMID 12028446
- [Background] Suzuki D, Yagame M, Kim Y, Sakai H, Mauer M. Renal in situ hybridization studies of extracellular matrix related molecules in type 1 diabetes mellitus. Nephron. 2002;92(3):564-72. doi: 10.1159/000064110. PMID 12372938
- [Background] Huang C, Kim Y, Caramori ML, Fish AJ, Rich SS, Miller ME, Russell GB, Mauer M. Cellular basis of diabetic nephropathy: II. The transforming growth factor-beta system and diabetic nephropathy lesions in type 1 diabetes. Diabetes. 2002 Dec;51(12):3577-81. doi: 10.2337/diabetes.51.12.3577. PMID 12453917
- [Background] Najafian B, Kim Y, Crosson JT, Mauer M. Atubular glomeruli and glomerulotubular junction abnormalities in diabetic nephropathy. J Am Soc Nephrol. 2003 Apr;14(4):908-17. doi: 10.1097/01.asn.0000057854.32413.81. PMID 12660325
- [Background] Caramori ML, Fioretto P, Mauer M. Low glomerular filtration rate in normoalbuminuric type 1 diabetic patients: an indicator of more advanced glomerular lesions. Diabetes. 2003 Apr;52(4):1036-40. doi: 10.2337/diabetes.52.4.1036. PMID 12663477
- [Background] Huang C, Kim Y, Caramori ML, Fish AJ, Rich SS, Miller ME, Russell GB, Mauer M. Cellular basis of diabetic nephropathy: III. In vitro GLUT1 mRNA expression and risk of diabetic nephropathy in type 1 diabetic patients. Diabetologia. 2004 Oct;47(10):1789-94. doi: 10.1007/s00125-004-1533-1. Epub 2004 Oct 22. PMID 15502921